CLINICAL TRIAL: NCT02767180
Title: Evaluation of an Intensive Care Specific Questionnaire for Patient-reported Outcome
Brief Title: Evaluation of an ICU-specific Questionnaire for Patient-reported Outcome Measures
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Stefan Lundin, Adjunct Professor, Sahlgrenska University Hospital
Other Study IDs: LUA-74200
Record Dates: First submitted 2016-04-28; First posted 2016-05-10 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Intensive Care Unit Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Critical care survivors: Former ICU-patients recruited six months to three years after discharge from the ICU
- Matched controls: Control patients who have not been critically ill, matched for age and sex.

SUMMARY:
An ICU-specific questionnaire for patient reported outcome measures (PROM) after critical care will be tested in a study of 650 patients recruited six months to three years after discharge from the ICU, and 150 controls who have not been critically ill, matched for age and sex. The questionnaire is sent by mail after an invitation letter followed by a phone call and returned in a pre-stamped envelope. It is then scanned and data imported digitally. Medical data from the ICU-stay can be added. Further analyses after comparison with the control population and item reduction will follow.

DETAILED DESCRIPTION:
ICU-patients were interviewed in a semi-structured way, providing detailed information on symptoms and difficulties in all areas of everyday life. The interviews were recorded, transcribed, and the issues were categorized into 13 hypothesised domains.All issues were then rephrased into questions, with care taken to maintain only one issue per question, and adequate scales for frequency, intensity and duration was used. The time frame is usually the last month. This intensive care specific questionnaire for patient reported outcome measures (PROM) after critical care will be tested in a study of 650 patients recruited six months to three years after discharge from the ICU, and 150 controls who have not been critically ill, matched for age and sex. The questionnaire is sent by mail after an invitation letter followed by a phone call and returned in a pre-stamped envelope. It is then scanned and data imported digitally. Medical data from the ICU-stay can be added. Further analyses after comparison with the control population and item reduction will follow.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated in an intensive care unit at Sahlgrenska University for more than 72 hours and survived are included between 6 months and tre years after discharge from ICU.
* Control persons from the Swedish Population Registry matched for sex and gender are also included.

Exclusion Criteria:

* Patient with acute neurological/neurosurgical conditions and/or anoxic/hypoxic brain damage

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients recruited six months to three years after discharge from the ICU, and 150 controls who have not been critically ill, matched for age and sex.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Patient reported outcome measured with an ICU-specific questionnaire | Six months to 3 years after intensive care
  An ICU-specific questionnaire will be used which has been developed from interviews of former ICU-patients

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Lundin, MD PhD, Principal Investigator — Dept of Anesthesia and Intensive Care, Sahlgrenska University Hospital, Gothenburg, Sweden
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Derived] Johannesson E, Malmgren J. Self-confidence as a mediator in the relationship between executive functioning and depression among ICU survivors: a latent variable analysis. Crit Care. 2024 Oct 26;28(1):345. doi: 10.1186/s13054-024-05136-2. PMID 39462425
- [Derived] Malmgren J, Lundin S, Waldenstrom AC, Rylander C, Johannesson E. Quality of life-related and non-quality of life-related issues in ICU survivors and non-ICU-treated controls: a multi-group exploratory factor analysis. Crit Care. 2024 Mar 29;28(1):102. doi: 10.1186/s13054-024-04890-7. PMID 38553749
- [Derived] Malmgren J, Waldenstrom AC, Rylander C, Johannesson E, Lundin S. Long-term health-related quality of life and burden of disease after intensive care: development of a patient-reported outcome measure. Crit Care. 2021 Feb 25;25(1):82. doi: 10.1186/s13054-021-03496-7. PMID 33632271